CLINICAL TRIAL: NCT03886181
Title: A Safety and Preliminary Effectiveness Study of Intratumoral Diffusing Alpha Radiation Emitters on Cutaneous, Mucosal and Superficial Soft Tissue Neoplasia
Brief Title: Alpha Radiation Emitters Device for the Treatment of Cutaneous, Mucosal and Superficial Soft Tissue Neoplasia (DaRT)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruitment and the site's resources to recruit patients
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-CMN-01
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Skin Cancer; Mucosal Neoplasm of Oral Cavity; Soft Tissue Neoplasm
Keywords: Squamous Cell Carcinoma; SCC; Skin Cancer; Skin metastasis; HNSCC; Carcinoma, Squamous; CMN; Basal cell carcinoma; Superficial sarcoma; Kaposi sarcoma; Alpha radiation; Cutaneous lesion; Tongue cancer; Lip cancer
MeSH Terms: conditions — Skin Neoplasms; Soft Tissue Neoplasms; Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Basal Cell; Sarcoma, Kaposi; Tongue Neoplasms; Lip Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for superficial cutaneous, mucosal or soft tissue neoplasia

DETAILED DESCRIPTION:
This will be a prospective, open label, single arm, controlled study, assessing the safety and efficacy of diffusing alpha emitters radiation therapy (DaRT) delivered through radioactive seeds inserted into the tumor.

This approach combines the advantages of local intratumoral irradiation of the tumor, as used in conventional brachytherapy, with the power of the alpha radiation emitting atoms, that will be introduced in quantities considerably lower than radiation therapy already used in patients.

Superficial lesions with histopathological confirmation of malignancy will be treated using DaRT seeds.

Reduction in tumor volume and evaluation the percent of necrotic tissue in the tumor 30-45 days after DaRT seeds insertion (15-30 days after seed removal) will be assessed. Safety will be assessed by the cumulative incidence, worst severity and frequency of adverse events (AEs) observed including the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histopathological confirmation of cutaneous and/or mucosal and/or superficial soft tissue malignant neoplasia.
* Subjects with a tumor size ≤ 5 centimeters in the longest diameter.
* Subjects' age is over 18 years old.
* Subjects' ECOG Performance Status Scale is < 2.
* Subjects' life expectancy is more than 6 months.
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test.
* Subjects are able and willing to sign an informed consent form.

Exclusion Criteria:

* Subject has a tumor with a maximal diameter > 5 centimeters.
* Subjects' ECOG Performance Status Scale is > 3.
* Subject has a tumor of Keratoacanthoma histology.
* Patients with moribund diseases, e.g., autoimmune diseases, vasculitis, etc.
* Patients under systemic immunosuppressive and/or corticosteroid treatment. Patients taking corticosteroid inhalers are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2024-10-13 (Actual); Study Completion 2024-10-13 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of the DaRT treatment | 5-7 weeks after DaRT seed insertion.
  The study primary objective is to evaluate the safety of the DaRT treatment in terms of incidence of device related Serious Adverse Events (SAE).

SECONDARY OUTCOMES:
Evaluation the effectiveness of the treatment. | Tumor volume will be measured during screening, 5 and 30-45 days post DaRT after treatment using CT.
  Evaluation on the effectiveness of the DaRT treatment, in terms of tumor volume reduction.

OTHER OUTCOMES:
Evaluate the effectiveness of the DaRT treatment, in terms of percent of necrotic | 15-30 days after removal of DaRT seeds.
  Evaluate the effectiveness of the DaRT treatment, in terms of percent of necrotic tissue present in the remaining tumor tissue surgically removed 15-30 days after removal of DaRT seeds.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Eibenschuz, MD, Principal Investigator — IFO S. Gallicano
Locations (1):
- IRCCS Istituto Dermatologico S. Gallicano, IFO - Istituti Fisioterapici Ospitalieri - Dermatologia Oncologica e Prevenzione, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No